CLINICAL TRIAL: NCT04885491
Title: An Open-Label, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of PDNO (Nitrosooxypropanol) Infusion in COVID-19 Patients With Acute Pulmonary Hypertension
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of PDNO Infusion in COVID-19 Patients With Acute Pulmonary Hypertension
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Since the availability of vaccines, a drastic drop in number of patients with increased PAP was observed and when the WHO re-categorized the COVID-19 pandemic from PHEIC to an "established and ongoing health issue" the study was withdrawn.
Sponsor: Attgeno AB (Industry)
Collaborators: Vinnova (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-PDNO-002
Record Dates: First submitted 2021-02-15; First posted 2021-05-13 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Hypertension; COVID-19
Keywords: Acute Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; COVID-19 | interventions — Sodium Chloride; 1-(nitrosooxy)propan-2-ol and 2-(nitrosooxy)propan-1-ol drug combination

STUDY DESIGN:
Intervention Model Description: Observational period with placebo treatment, followed by treatment with PDNO.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with PDNO (Experimental): Placebo treatment administered during the 120-minute observation period, followed by PDNO infusion. PDNO administered as an i.v. infusion of 5-15 minutes, respectively, for the increased planned dose titration steps: 3, 10 and thereafter steps of max 10 nmol/kg/min until the target effect on the mean pulmonary arterial pressure/pulmonary vascular resistance (MPAP/PVR) or a maximal dose of 120 nmol/kg/min is reached.
  After 4 patients have been treated, the internal safety review committee (iSRC) will decide if the start dose will be increased. The new start dose could be in the interval 1 to 5 nmol/kg/min.
  Interventions: Drug: Sodium chloride (placebo); Drug: PDNO

INTERVENTIONS:
Drug: Sodium chloride (placebo) — Placebo (NaCl, commercially available dilution solution for parenteral use, 9 mg/mL)
  Other Names: NaCl
Drug: PDNO — PDNO consists of propylene glycol (1,2-propanediol, PD) chemically combined with NO (to be donated). The drug substance is formulated as an inherent mixture of 4 structure analogues. The mixture consists of an equilibrium of the 2 regioisomers 1-(nitrosooxy) propan-2-ol and 2-(nitrosooxy) propan-1-ol. In addition, each regioisomer is a racemic mixture.
  Other Names: Nitrosooxypropanol

SUMMARY:
This is an open-label, multicentre study evaluating the effect, safety and tolerability of the two regioisomers 1-(nitrosooxy)propan-2-ol and 2-(nitrosooxy)propan-1-ol (PDNO) infusion given to COVID-19 patients with acute pulmonary hypertension (aPH) and/or acute cor pulmonale (ACP).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willing to sign an ICF
* Male and female patients at least 18 years of age
* Diagnosed with COVID-19 at admission to the ICU
* Diagnosed with echocardiographic signs of pulmonary artery systolic pressure (PASP) > 40 mmHg

Exclusion Criteria:

* History of chronic pulmonary hypertension (PH), as judged by the Investigator at screening
* Known New York Heart Association (NYHA) Functional Class III or IV symptoms
* Left heart failure with ejection fraction (EF) < 35%
* Acute coronary syndrome
* Body Mass Index (BMI) > 45 kg/m^2
* Estimated glomerular filtration rate (eGFR) < 30 mL/min
* MetHb > 3%
* PCO2 > 7
* Indication of liver disease, defined by serum levels of either alanine aminotransferase (ALT), aspartate aminotransferase (AST) or alkaline phosphatase (ALP) above 3 x upper limit of normal (ULN) at screening
* Haemoglobin < 80 g/dL
* Thrombocytopenia (platelet count < 80000/mm^3)
* Prothrombin time International ratio (INR) > 1.4
* Pregnancy, or a positive pregnancy test
* Ongoing daily treatment the last 3 days with non-steroidal anti-inflammatory drugs
* Known active malignancy within the past 3 years
* History of allergy/hypersensitivity to PD or ongoing allergy/hypersensitivity or history of hypersensitivity to drugs with a similar chemical structure or class to PDNO
* History of any other clinically significant disease or disorder
* Participation in any interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in MPAP and calculated PVR measured with PAC, at target dose after up-titration and 10 minutes after steady state. | During 24 hours
  Mean pulmonary arterial pressure (MPAP) and pulmonary vascular resistance (PVR), as measured with a pulmonary artery catheter (PAC).

SECONDARY OUTCOMES:
Safety and tolerability of PDNO in patients with COVID-19, as measured by incidence of treatment-emergent AEs, SAEs, and AESI. | Through study completion (i.e., Day 30)
  * Treatment-emergent adverse events (AEs)
  * Treatment-emergent serious AEs (SAEs)
  * Treatment-emergent AEs of special interest (AESI)
Safety and tolerability of PDNO in patients with COVID-19, as measured by incidence of treatment-emergent changes in vital signs, ECG abnormalities, and laboratory abnormalities. | From baseline until Day 7
  * Treatment-emergent changes in vital signs (blood pressure, pulse, oxygen saturation, respiratory frequency, body temperature)
  * Treatment-emergent electrocardiogram (ECG) abnormalities
  * Treatment-emergent laboratory abnormalities
Number of participants with the following clinical outcome (dead, intubated at the intensive care unit [ICU], non-intubated at the ICU, discharged from ICU to other hospital care or discharged to home). | At Days 7, 14, 21, and 30.
Time to obtain first negative upper respiratory tract sample in the SARS-CoV-2-rt-PCR assay | From Day 1 to Day 14
Change in troponin I/T and BNP/NT-proBNP | From end of PDNO infusion to Day 7.
Change in the ratio PVR/SVR | During 24 hours
  Pulmonary vascular resistance (PVR) and systemic vascular resistance (SVR) will be calculated from the obtained values according to the following formulas:
  PVR= (mean pulmonary arterial pressure [MPAP] - pulmonary capillary wedge pressure [PCWP])/cardiac output (CO) SVR= (mean arterial pressure [MAP] - central venous pressure [CVP])/CO
  Ratio of PVR to SVR = PVR/SVR

OTHER OUTCOMES:
Levels of SARS-CoV-2 virus in plasma and sputum/tracheal secretion | From Day 1 to Day 2
Collection of plasma for future analysis of biomarkers such as nitrite and nitrate in plasma (µM) | From Day 1 to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Kemi, PhD, Study Director — Attgeno AB
Locations (2):
- Sweden (2):
  - Danderyd Hospital, Danderyd
  - Örebro University Hospital, Örebro

IPD SHARING:
Plan to Share IPD: No